CLINICAL TRIAL: NCT05325684
Title: Efficacy and Safety of PD-L1 Inhibitor in Patients With Advanced Solid Tumors Beyond Lung Cancer: a PhaseⅠB Clinical Study
Brief Title: PD-L1 Inhibitor Rechallenge After PD-1 Immunotherapy for Patients With Solid Tumor Beyond Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, zhangxiaochun, director, The Affiliated Hospital of Qingdao University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDL1-BEY-LUNG
Record Dates: First submitted 2022-03-31; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Efficacy; Safety
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-L1 rechallenge (Experimental)
  Interventions: Drug: PD-L1 inhibitor

INTERVENTIONS:
Drug: PD-L1 inhibitor — Enrolled patients received durvalumab/ Atezolizumab plus chemotherapy or target therapy treatment (durvalumab,1000mg，iv, d1, 21day as a cycle; Atezolizumab,1200mg iv, d1, 21day as a cycle.)

SUMMARY:
Anti-PD-L1 immune checkpoint inhibitor, is approved for the treatment of patients with unresectable, Stage III NSCLC whose disease has not progressed following concurrent platinum-based chemotherapy and radiation therapy, or as first-line treatment of patients with ES-SCLC in combination with etoposide and either carboplatin or cisplatin in China. The clinical data regarding the PD-L1 inhibitor in other solid tumors are limited.Investigators would observe and analyze the effectiveness and safety of PD-L1 inhibitor for patients with advanced - solid tumors beyond lung cancer after muti-line therapy to explore the synergistic effect of PD-L1 inhibitor rechallenge after PD-1immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Ability to comply with protocol
* Aged ≥ 18 years
* Histologically documented advanced solid tumor beyond lung cancer
* Disease progression during or following at least one line treatment containing PD-1 immunotherapy.
* Measurable disease, as defined by RECIST v1.1
* ECOG performance status of 0 or 1
* Life expectancy ≥ 12 weeks
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment:

ANC ≥ 1.5 × 109/L (without granulocyte colony-stimulating factor support within 2 weeks of laboratory test used to determine eligibility) WBC counts > 2.5 × 109/L and < 15 × 109/L Lymphocyte count ≥ 0.5 × 109/L Serum albumin ≥ 2.5 g/dL Platelet count ≥ 100 × 109/L (without transfusion within 2 weeks of laboratory test used to determine eligibility) Hemoglobin ≥ 9.0 g/dL Patients may be transfused or receive erythropoietic treatment to meet this criterion.

Liver function tests meeting one of the following criteria:

AST or ALT ≤ 2.5 × upper limit of normal (ULN), with alkaline phosphatase

≤ 2.5 × ULN or AST and ALT ≤ 1.5 × ULN in conjunction with alkaline phosphatase > 2.5 × ULN Serum bilirubin ≤ 1.5 × ULN Patients with known Gilbert's disease who have serum bilirubin level ≤ 3 × ULN may be enrolled. INR and aPTT ≤ 1.5 × ULN This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose for at least 1 week prior to randomization. Creatinine clearance ≥ 30 mL/min Cockcroft-Gault, Chronic Kidney Disease Epidemiology Collaboration, or Modification of Diet in Renal Disease formulas may be used for creatinine clearance calculation. Note that 24-hour urine collection is not required but is allowed.

Exclusion Criteria:

* Active or untreated CNS metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled hypertension
* Autoimmune disease
* Had undergone a serious anaphylactic reaction in previous immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
DCR | At the end of Cycle 3 (each cycle is 21 days)".
  Disease Control Rate
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  progression-free survival

SECONDARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months
  overall survival
AE | hrough study completion, an average of 1 year
  adverse event caused by the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Zhang, Prof, Principal Investigator — The Affiliated Hospital of Qingdao University